CLINICAL TRIAL: NCT04530175
Title: Modeling of Regional Citrate Anticoagulation With a Dialysate Containing Calcium in Intermittent Hemodialysis
Brief Title: Modeling of Regional Citrate Anticoagulation With a Dialysate Containing Calcium in Intermittent Hemodialysis (MARC)
Acronym: MARC
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RBHP 2020 ANIORT; 2020-A01359-30 (Other: ANSM)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: End Stage Renal Disease
Keywords: hemodialysis; modeling; Citrate anticoagulation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with hemodialysis: patient treated with intermittent hemodialysis for chronic renal failure
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — 2 blood samples will be taken from the blood circuit 1 hour after the start of the hemodialysis session by the nurse in charge of the patient.

SUMMARY:
The primary purpose of this study is to validate a mathematical modeling of treatment by intermittent hemodialysis using regional citrate anticoagulation with a dialysate containing calcium

DETAILED DESCRIPTION:
The only visit to the study will be carried out during a usual dialysis session in the intensive care unit of Clermont-Ferrand University Hospital. In addition to the usual care, 2 blood samples will be taken from the blood circuit 1 hour after the start of the hemodialysis session by the nurse in charge of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Major patient;
* Man or woman ;
* Treated with intermittent hemodialysis for chronic renal failure;
* In whom intermittent hemodialysis with citrate solution for regional anticoagulation is indicated;
* Affiliated with a social security scheme;
* Having given a signed agreement after detailed explanation of the protocol on the basis of the information sheet and likely to comply with it

Exclusion Criteria:

* Severe hepato-cellular insufficiency (PT <50%, INR> 1.5 without anticoagulant);
* Hemoglobin level <7 g / dL
* Presenting a psychiatric pathology or cognitive impairment rendering him unable to give informed consent;
* Persons under guardianship, curatorship, deprived of liberty or safeguard of justice
* Pregnant or breastfeeding women
* Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with intermittent hemodialysis for chronic renal failure, at university hospital of Clermont-Ferrand
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Ionized calcium level | day 0
  measured at dialyzer inlet, in mmol/L
Total calcium level | day 0
  measured at dialyzer inlet, in mmol/L
Total citratemia | day 0
  measured at dialyzer inlet, in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Julien Aniort, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France